CLINICAL TRIAL: NCT04940156
Title: Comparison of the Performance of Implantable Cardiac Monitors and Cardiac Implantable Electronic Devices in Detecting Atrial Fibrillation
Brief Title: Comparison of the Performance of ICM and CIED in Detecting AF
Acronym: ID-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment to study was insufficient. This was despite extending the recruitment period. Decision taken to terminate study due to lack of recruitment.
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14558
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
Keywords: Confirm Rx; Reveal LINQ
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients implanted with the Abbott Confirm Rx ICM (Other): Patient with cardiac implantable electronic devices with an atrial lead will have Confirm Rx Implantable Cardiac Monitor injected in the anterior chest wall.
  Interventions: Device: Confirm Rx (Implantable Cardiac Monitor)
- Patients implanted with the Medtronic LINQ ICM (Other): Patient with cardiac implantable electronic devices with an atrial lead will have LINQ Implantable Cardiac Monitor injected in the anterior chest wall.
  Interventions: Device: Reveal LINQ (Implantable Cardiac Monitor)

INTERVENTIONS:
Device: Confirm Rx (Implantable Cardiac Monitor) — Confirm Rx implanted in patients with atrial fibrillation detected on their cardiac implantable electronic device (CIED)
  Arms: Patients implanted with the Abbott Confirm Rx ICM
Device: Reveal LINQ (Implantable Cardiac Monitor) — Reveal LINQ implanted in patients with atrial fibrillation detected on their cardiac implantable electronic device (CIED)
  Arms: Patients implanted with the Medtronic LINQ ICM

SUMMARY:
The aim of this project is to study the performance of the two most commonly used Implantable Cardiac Monitors in detecting AF episodes and explore how the new connectivity can empower patients and improve patient care.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common abnormal heart rhythm disturbance, affecting 1-2 million people in the UK. The irregular heartbeat caused by AF can make the heart pump blood less efficiently. As a result, AF significantly increases the risk of having a stroke, heart failure and dementia. However, a significantly proportion of people have no symptoms, and they may be only found to be in AF after having a stroke. Therefore, diagnosis largely relies on accurate electrocardiogram (ECG) monitoring.

AF episodes can be unpredictable and easily missed unless continuous ECG monitoring is undertaken. Pacemakers can continuously record the heart's electrical activity and detect AF with a high degree of confidence. However, they are invasive and rely on electrical wires implanted inside the heart, and hence less suited to be used as primary monitoring devices. To overcome these difficulties, implantable cardiac monitors (ICM) have been designed to be placed under the skin.

The new generation of ICMs can now be injected under the skin. Moreover, they connect with the patient's smartphone and transmit recordings. Despite these significant improvements, their ability to reliably capture AF has never been tested against pacemakers.

The aim of this project is to study the performance of the two commonly used ICMs in detecting AF episodes and explore how the new connectivity can empower patients and improve patient care. The investigators plan to inject an ICM in 30 patients with AF and pre-existing pacemaker. After a period of 6 months, the investigators will compare how many episodes were detected in each device. With the information collected the investigators will try to understand the pitfalls in the current technology and develop strategies to improve it.

Accurate, minimally invasive long-term ECG monitor can have far reaching benefits for patients, both in routine clinical practice and research.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female.
* Aged 18 years or above.
* History of paroxysmal and persistent AF.
* Dual-chamber pacemaker, Implantable cardioverter defibrillator (ICD) or cardiac resynchronisation therapy (CRT) device with a functioning atrial lead, able to record electrograms and remote monitoring.

Exclusion Criteria:

* Diagnosis of permanent AF.
* Contra-indications for implantable cardiac monitor.
* Unable to comply with the follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Betts, MD FRCP, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Confirm Rx: Patient with cardiac implantable electronic devices with an atrial lead will have Confirm Rx Implantable Cardiac Monitor injected in the anterior chest wall.
  Confirm Rx (Implantable Cardiac Monitor): Confirm Rx implanted in patients with atrial fibrillation detected on their cardiac implantable electronic device (CIED)
- LINQ: Patient with cardiac implantable electronic devices with an atrial lead will have LINQ Implantable Cardiac Monitor injected in the anterior chest wall.
  Reveal LINQ (Implantable Cardiac Monitor): Reveal LINQ implanted in patients with atrial fibrillation detected on their cardiac implantable electronic device (CIED)
Period: Overall Study
Arm/Group | Confirm Rx | LINQ
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients recruited from Cardiac clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Confirm Rx | LINQ | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5 | 1 | 6
Count of participants [Count of Participants; unit: Participants] | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Performance of Confirm Rx ICM and Reveal LINQ ICM in Detecting AF Episodes in Comparison to CIED
Description: To assess the performance of the Confirm Rx™ ICM and Reveal LINQ™ ICM in detecting clinically significant AF episodes (episodes longer than 6 minutes) in comparison to CIED (gold standard). Confirm Rx and Reveal LINQ™ ICM sensitivity, specificity, positive predictive value and negative predictive value will be calculated for AF episodes longer than 6 minutes.
Time Frame: During follow-up (6 months)
Population: Data were not collected.
Arm/Group | Confirm Rx | LINQ
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Comparison of Changes in R-wave Amplitude Following Implantation in Both ICMs.
Description: A comparison will be made between the percentage of change in R-wave amplitudes between both ICMs.
Time Frame: During follow-up (6 months)
Population: Data were not collected.
Arm/Group | Confirm Rx | LINQ
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Compare the Transmission Success Rate of Both Devices.
Description: The percentage of successful transmission in both ICMs will be calculated.
Time Frame: During follow-up (6 months)
Population: Data were not collected.
Arm/Group | Confirm Rx | LINQ
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Compare the Number of Patient-activated Recordings That Contains Symptoms.
Description: The percentage of patient-activated recordings with symptoms attributed to those episodes will be calculated.
Time Frame: During follow-up (6 months)
Population: Data were not collected.
Arm/Group | Confirm Rx | LINQ
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Confirm Rx | LINQ
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 0/5 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT04940156/Prot_SAP_000.pdf